CLINICAL TRIAL: NCT03043911
Title: Improved Patient Safety Through Continuous Bi-channel Respiratory Rate and Oxygen Saturation Monitoring With Masimo Patient SafetyNet
Brief Title: Improved Patient Safety Through Continuous Bi-channel RR and SpO2 Monitoring With Masimo Patient SafetyNet
Acronym: SafetyNet
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Baylor Research Institute (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 014-293
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Signs and Symptoms, Respiratory
Keywords: early detection; respiratory events; sepsis
MeSH Terms: conditions — Signs and Symptoms, Respiratory; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigator intend to perform an observational study, by adding Respiratory Rate monitoring to an already existing Patient SafetyNet system with SpO2 (Oxygen Saturation) and PR (Pulse Rate) monitoring. RRa will be blinded to the clinicians and all RRa alarms will be deactivated. Retrospective analysis of the observational data collected will be utilized to evaluate the potential benefits of additional continuous respiratory rate monitoring.

DETAILED DESCRIPTION:
Addition of acoustic respiratory rate monitoring to an already existing standard of care patient surveillance system that includes oxygen saturation and heart rate monitoring by pulse oximetry will result in earlier and more sensitive detection of respiratory events and possibly early stages of developing sepsis in a post-surgical/orthopedic study population.

An observational study with RRa is an additional blinded parameter to the already existing standard of care monitoring with SpO2 and PR on one post-surgical floor, (includes Trauma and orthopedic patients), where patients receive opioids for pain management. 300 consecutive patients will be enrolled and monitored with RRa for at least the first 24hours post-surgery, after discharge from the Recovery Room, & upon admission to the Surgical floor.

ELIGIBILITY:
Inclusion Criteria:

* • Adult 18yrs of age or older

  * Post-surgical patient receiving opioid pain medication

Exclusion Criteria:

* • Refusal of optical finger sensor and/or acoustic respiratory rate neck sensor placement

  * Finger or skin abnormalities at sensor sites
  * Expected opioid therapy duration less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients to be admitted to the general post surgical floor who meet the inclusion and exclusion criteria will be enrolled after signing the study consent form.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Improved sensitivity of RRa by detecting the number and the incidence rate of respiratory depression events | with in 24 hours post surgery

SECONDARY OUTCOMES:
Time period between detection of first early symptoms of developing sepsis with RRa, PR and SpO2 monitoring compared to the first clinical diagnosis of developing sepsis. | with in 24 hours post surgery